CLINICAL TRIAL: NCT06072534
Title: Evaluation of Effectiveness of Two Different Doses of Mivacurium in Modified Rapid Sequence Intubation for Emergency Surgery ,Prospective Randomized Double Blind Study
Brief Title: Evaluation of Effectiveness of Two Different Doses of Mivacurium in Rapid Sequence Intubation
Acronym: RSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ismail Mohamed Abdelgawad Ahmed, DOCTOR, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: mivacurium in RSI
Record Dates: First submitted 2023-09-03; First posted 2023-10-10 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Emergencies
Keywords: mivacurium; rapid sequence intubation; emergency surgery
MeSH Terms: conditions — Emergencies | interventions — Mivacurium

STUDY DESIGN:
Intervention Model Description: prospective randomized double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Miva 3 (Active Comparator): "Mivacurium chloride" ("Mivacron®") 0.3 mg/kg 3 times effective dose (ED) 95 iv during induction recording intubation condition during rapid sequence intubation within 90 sc monitoring hemodynamic changes during intubation ,time to recover to T1
  Interventions: Drug: "Mivacurium Chloride"
- Miva 4 (Active Comparator): "Mivacurium chloride" ("Mivacron®") 0.4 mg/kg 4 times effective dose (ED) 95 iv during induction
  recording intubation condition during rapid sequence intubation within 90 sc monitoring hemodynamic changes during intubation,time to recover to T1
  Interventions: Drug: "Mivacurium Chloride"

INTERVENTIONS:
Drug: "Mivacurium Chloride" — emergence modified sequence intubation
  Other Names: "Mivacron®"

SUMMARY:
Mivacurium can be considered as an optimal choice for muscle relaxation in short duration surgeries, as butyrylcholinesterase can rapidly and reliably degrade this benzylisoquinoline muscle relaxant in vivo. However the histamine release related to a rapid high-dose injection, unsatisfactory intubation conditions and unexpected delay in recovery in patients may be encountered with butyrylcholinesterase deficiency

DETAILED DESCRIPTION:
Intubation in emergency and full stomach patients stands as a challenge in anaesthesia. Rapid sequence induction (RSI) is the key player technique in avoiding gastric contents aspiration risk. Non-depolarizing neuromuscular blocking agents as mivacurium are of clinical significance in the anesthetic management of patient. Mivacurium has been has been preferred in situations who necessitating hemodynamic solidity all over the surgery, as only transient tachycardia and hypotension were recorded

Aim of work Using high doses of mivacurium can provide accepted condition of emergency intubation within favorable time - monitoring hemodynamics changes during and after intubation, time of recovery from high doses of muscle relaxant

ELIGIBILITY:
Inclusion Criteria:

* 20-60 year old patients.
* American society of anaesthesia (ASA) 1 and 2.
* Emergency surgery.

Exclusion Criteria:

* Refusal.
* allergy.
* neuromuscular disease.
* Suspected desaturation.
* Severe cardiac disease.
* Severe pulmonary disease.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Intubation conditions during RSI. | 3 months
  Jaw relaxation or ease blade insertion was graded as easy (3), moderate (2), difficult (1) and impossible (0).
  Vocal cord positions were ranked as abducted (3), moving (2), closing (1) and closed (0). Response to intubation was graded as no movement (3), slight diaphragmatic movement (2), mild coughing (1) and severe coughing or bucking (0).
  The total scores of the three variables were rated as excellent (8-9), good (6-7), fair (3-5) and poor (0-2).
  Good and excellent intubating conditions were considered 'clinically acceptable'.

SECONDARY OUTCOMES:
change in heart rate beat/minute: | 12 weeks
  * pre-induction.
  * every 1 minute for 5 minutes after intubation
change in mean arterial bood pressure (MAP) mmHg/minute: | 12 weeks
  * pre-induction.
  * every 1 minute for 5 minutes after intubating
time/minute to T1 recovery monitoring | 12 weeks
  by train-of-four (TOF) every 5 minutes until one twitch of TOF

CONTACTS AND LOCATIONS:
Overall Officials: ismail m ahmed, professor, Principal Investigator — Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: No
the patient will be coded

REFERENCES:
- [Background] Savarese JJ, Ali HH, Basta SJ, Embree PB, Scott RP, Sunder N, Weakly JN, Wastila WB, el-Sayad HA. The clinical neuromuscular pharmacology of mivacurium chloride (BW B1090U). A short-acting nondepolarizing ester neuromuscular blocking drug. Anesthesiology. 1988 May;68(5):723-32. doi: 10.1097/00000542-198805000-00010. PMID 2967039
- [Background] Ostergaard D, Viby-Mogensen J, Rasmussen SN, Gatke MR, Pedersen NA, Skovgaard LT. Pharmacokinetics and pharmacodynamics of mivacurium in patients phenotypically heterozygous for the usual and atypical plasma cholinesterase variants (UA). Acta Anaesthesiol Scand. 2003 Nov;47(10):1219-25. doi: 10.1046/j.1399-6576.2003.00243.x. PMID 14616318
- [Background] Plaud B, Marty J, Debaene B, Meistelman C, Pellissier D, LePage JY, Feiss P, Scherpereel P, Bouverne MN, Fosse S. The cardiovascular effects of mivacurium in hypertensive patients. Anesth Analg. 2002 Aug;95(2):379-84, table of contents. doi: 10.1097/00000539-200208000-00025. PMID 12145055
- [Background] Cooper R, Mirakhur RK, Clarke RS, Boules Z. Comparison of intubating conditions after administration of Org 9246 (rocuronium) and suxamethonium. Br J Anaesth. 1992 Sep;69(3):269-73. doi: 10.1093/bja/69.3.269. PMID 1389845